CLINICAL TRIAL: NCT02368535
Title: A Decade of Safon Rounds: Interdisciplinary Daily Rounding as a Method of Improving Teamwork in an Academic, Tertiary Care Labor and Delivery Unit
Brief Title: Improving Teamwork in an Academic, Tertiary Care Labor and Delivery Unit
Acronym: SAFON
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Vice-Chair, Faculty Development and Education, Brigham and Women's Hospital
Other Study IDs: SAFON STUDY
Record Dates: First submitted 2015-02-06; First posted 2015-02-23 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Interdisciplinary Communication
Keywords: teamwork
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey — 25-item questionnaire on pereception of interdisciplinary rounds

SUMMARY:
The investigators wanted to determine if the establishment of interdisciplinary rounds has made meaningful changes in the perceptions of teamwork and communication.

The purpose of this study is to determine if the establishment of interdisciplinary daily rounding has improved teamwork in an academic, tertiary care labor and delivery unit.

DETAILED DESCRIPTION:
Failures in teamwork and communication are among the leading cases of sentinel and adverse obstetric events. Multidisciplinary approaches and communication could improve patients outcomes. In 2003, leaders from the department of obstetrics, anesthesia and nursing decided to institute interdisciplinary rounds as a method of improving team communication. Obstetricians, Anesthesiologists, Nurses, Perinatologists, Administrative Assistants, Consultants, and Neonatologists participate in the rounds. The investigators wanted to determine if the establishment of interdisciplinary rounds has made meaningful changes in the perceptions of teamwork and communication.

The purpose of this study is to determine if the establishment of interdisciplinary daily rounding has improved teamwork in an academic, tertiary care labor and delivery unit.

ELIGIBILITY:
Inclusion Criteria:

* Working at L&D at Brigham and Women's and participating in daily rounds

Exclusion Criteria:

* subject's refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Staff working at Brigham and Women's Hospital Labor and Delivery Suite
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Perception of Teamwork Elements Present in Interdisciplinary Rounds - Total Response Scores | Individual Participation-10 min; Study Completion within 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Tsen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States